CLINICAL TRIAL: NCT01169649
Title: A Phase II Clinical and Translational Study of MK-2206 in Patients With Metastatic Neuroendocrine Tumors (NET)
Brief Title: Study of MK-2206 in Patients With Metastatic Neuroendocrine Tumors (NET)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-067
Record Dates: First submitted 2010-07-21; First posted 2010-07-26 (Estimated); Results first posted 2016-02-18 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-01

CONDITIONS: PANCREAS; Neuroendocrine
Keywords: MK-2206; Neuroendocrine Tumors; 10-067
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — MK 2206

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- islet cell carcinomas and carcinoid tumors (Experimental): This is an open label phase II study of MK-2206 administered to patients with metastatic neuroendocrine tumors.
  Interventions: Drug: MK-2206

INTERVENTIONS:
Drug: MK-2206 — MK-2206 will be given orally 200 mg qw as given in the prior Ph1 clinical trial that demonstrated safety, tolerability and adequate PK/PD values at this dose. Follow-up imaging scans will be performed every 12 weeks to evaluate response. Patients must take MK-2206 orally at least 2 hours before or 2 hours after food or a meal.

SUMMARY:
The purpose of this study is to test a new drug called MK-2206. This study is a phase II study. In cancer studies, a phase II study is to find out what effects, good and/or bad, a new treatment has against a certain type of cancer.

MK-2206 is an oral medication known as a targeted therapy. By attaching to the target, we hope that MK-2206 may stop the cancer cells from further growth and dividing. This study will help find out if MK-2206 is a helpful drug when taken in patients with neuroendocrine tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed moderately to well differentiated metastatic or unresectable carcinoid or islet cell tumors.
* Patient has at least one measurable lesion greater than or equal to 20 mm on CT or MRI imaging.
* Patients who are on therapy with a somatostatin analog are eligible for entry but must be on a stable dose for at least 3 months with no evidence of tumor shrinkage during that time period.
* Patient ≥18 years of age on the day of signing informed consent.
* Patient has performance status 0-1 on the ECOG Performance Scale.
* Patient has adequate organ function as indicated by the following laboratory values:
* Absolute Neutrophil Count (ANC)≥1,500/mcL
* Platelets ≥100,000/mcL
* Hemoglobin ≥9 g/dL
* Serum Creatinine ≤2 times the upper limit of normal (ULN)/ OR calculated CrCl ≥60 mL/min (patients with creatinine levels ≥2 times the ULN only). Patient may not be on dialysis
* Serum total bilirubin ≤1.5 times the ULN
* AST (SGOT) and ALT (SGPT) ≤5 times the ULN
* HgbA1c ≤ 8%
* Fasting Glucose ≤120 mg/dl
* Creatinine clearance should be calculated by the Cockcroft-Gault method.Fasting is defined as at least 4 hours without oral intake.
* Patient has voluntarily agreed to participate by giving written informed consent.
* Previous local therapy (e.g. chemoembolization or bland embolization) is allowed if completed > 6 weeks or 5X half-life prior to study entry. For patients who received local therapy prior to study entry, there must be either documented growth of measurable disease within the embolization field or outside of the embolization field, or both, prior to study entry if the area of the embolization field was the only site of measurable disease.
* Previous chemotherapy, radiotherapy, and/or biologic therapy, including investigational agents, is/are allowed if completed > 4 weeks prior to study entry (>6 weeks if last regimen contained bevacizumab, BCNU or mitomycin C, and > 6 weeks from last dose of radiation therapy or radiopharmaceutical.
* Patients must not have disease that is currently amenable to curative surgery. Prior surgery is allowed no less than 6 weeks prior to study entry.
* Patients with diabetes mellitus are eligible for study entry but must have controlled diabetes as defined by hemoglobin A1c <8.0% within 2 weeks of initiation of protocol therapy.

Exclusion Criteria:

* Patient has toxicities from prior therapies that have not resolved to grade 1 or grade 0.
* Patient has known active CNS metastases and/or carcinomatous meningitis are excluded. However, patients with CNS metastases who have completed a course of therapy would be eligible for the study provided they are clinically stable for 1 month prior to entry as defined as: (1) no evidence of new or enlarging CNS metastasis (2) off steroids that are used to minimize surrounding brain edema.
* Patient has an active malignancy of metastatic potential other than the known carcinoid or islet cell tumor, for the past 3 years.
* Patient has a known hypersensitivity to the components of study drug (MK-2206) or its analogs that is not treatable by premedication with antihistamines and steroids.
* Patient has a condition, including but not limited to
* symptomatic congestive heart failure
* unstable angina pectoris
* serious cardiac arrhythmia
* history or current evidence of a myocardial infarction during the last 6 months, and/or a current ECG tracing that is abnormal in the opinion of the treating investigator
* QTc prolongation >450 msec (Bazett's formula)
* Patient with evidence of clinically significant bradycardia (HR <50), or a history of clinically significant bradyarrhythmias such as sick sinus syndrome, 2nd degree AV block (Mobitz Type 2).
* Patient with uncontrolled hypertension (i.e., 160/90 mHg SiBP). Patients who are controlled on antihypertensive medication will be allowed to enter the study.
* Patient at significant risk for hypokalemia (e.g., patients on high dose diuretics, or with recurrent diarrhea)
* Patient is a known diabetic who is poorly controlled (HBAc>8%)
* Patient has a history or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
* Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Patient is, at the time of signing informed consent, a regular user (including -recreational use‖) of any illicit drugs or had a recent history (within the last year) of drug or alcohol abuse.
* Patient is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.
* Patient is known to be Human Immunodeficiency Virus (HIV)-positive
* Patient has known history of Hepatitis C or active Hepatitis A or B.
* Patient has symptomatic ascites or pleural effusion. A patient who is clinically stable following treatment for these conditions is eligible.
* Patient has prior treatment with an mTOR inhibitor such as afinitor, sirolimus, or temsirolimus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Reidy-Lagunes, MD,MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-2206 in Patients With Metastatic Neuroendocrine Tumors: This is an open label phase II study of MK-2206 administered to patients with metastatic neuroendocrine tumors.
Period: Overall Study
Arm/Group | MK-2206 in Patients With Metastatic Neuroendocrine Tumors
Started | 11
Completed | 8
Not Completed | 3
Not completed — Patient Not Treated | 3

BASELINE CHARACTERISTICS:
Arm/Group | MK-2206 in Patients With Metastatic Neuroendocrine Tumors
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Response.
Description: Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: every 12 weeks
Measure: Number; unit: participants
Arm/Group | MK-2206 in Patients With Metastatic Neuroendocrine Tumors
Number analyzed (Participants) | 8
participants
  Stable Disease | 6
  Progression of Disease | 2

ADVERSE EVENTS:
Arm/Group | MK-2206 in Patients With Metastatic Neuroendocrine Tumors
Serious Adverse Events (participants affected / at risk) | 4/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-2206 in Patients With Metastatic Neuroendocrine Tumors (N=8)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-2206 in Patients With Metastatic Neuroendocrine Tumors (N=8)
Alanine aminotransferase increased (Blood and lymphatic system disorders) | 2 (2)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 3 (3)
Anorexia (General disorders) | 1 (1)
Aspartate aminotransferase increased (Blood and lymphatic system disorders) | 2 (2)
Blood bilirubin increased (Metabolism and nutrition disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Lipase increased (Metabolism and nutrition disorders) | 1 (1)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4)
Serum amylase increased (Metabolism and nutrition disorders) | 1 (1)
White blood cell decreased (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes